CLINICAL TRIAL: NCT00837954
Title: Randomized, Controlled, Prospective Trial to Evaluate the Hemostatic Effect of Lyostypt® Versus Surgicel® in Arterial Bypass Anastomosis
Brief Title: Trial to Evaluate the Hemostatic Effect of Lyostypt® Versus Surgicel® in Arterial Bypass Anastomosis
Acronym: COBBANA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAG-G-H-0803
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Peripheral Vascular Diseases; Hemostasis
Keywords: PTFE Graft; Suture Hole Bleeding; Hemostasis
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Surgicel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): distal Anastomosis Lyostypt®, proximal Anastomosis Surgicel®
  Interventions: Device: Lyostypt® AND Surgicel®
- 2 (Active Comparator): distal Anastomosis Surgicel®, proximal Anastomosis Lyostypt®
  Interventions: Device: Lyostypt® AND Surgicel®
- 3 (Active Comparator): distal and proximal Anastomosis Lyostypt®
  Interventions: Device: Lyostypt®
- 4 (Active Comparator): distal and proximal Anastomosis Surgicel®
  Interventions: Procedure: Surgicel®

INTERVENTIONS:
Device: Lyostypt® AND Surgicel® — The investigational products are the hemostats Lyostypt® and Surgicel® (=Tabotamp® ). Lyostypt® will be provided in the size 5cm x 8cm, Surgicel® will be provided in the size 5cm x 7,5cm. The devices will be cut into half.
  Lyostypt® is an absorbable wet-stable collagen compress made of collagen fibrils of bovine origin. Collagen leads to thrombocyte adhesion and to activation of coagulation factor XII.
  Surgicel® absorbable Haemostat is a sterile absorbable knitted fabric prepared by the controlled oxidation of regenerated cellulose. After Surgicel® has been saturated with blood, it swells into a brownish or black gelatinous mass which aids in the formation of a clot, thereby serving as a haemostatic adjunct in the control of local haemorrhage.
  Other Names: Lyostypt®; Surgicel®
  Arms: 1; 2
Device: Lyostypt® — The investigational product is the hemostat Lyostypt®. Lyostypt® will be provided in the size 5cm x 8cm. The devices will be cut into half.
  Lyostypt® is an absorbable wet-stable collagen compress made of collagen fibrils of bovine origin. Collagen leads to thrombocyte adhesion and to activation of coagulation factor XII.
  Arms: 3
Procedure: Surgicel® — The investigational product is the hemostat Surgicel® (=Tabotamp® ). Surgicel® will be provided in the size 5cm x 7,5cm. The devices will be cut into half.
  Surgicel® absorbable Haemostat is a sterile absorbable knitted fabric prepared by the controlled oxidation of regenerated cellulose. After Surgicel® has been saturated with blood, it swells into a brownish or black gelatinous mass which aids in the formation of a clot, thereby serving as a haemostatic adjunct in the control of local haemorrhage.
  Arms: 4

SUMMARY:
The purpose of this trial is to demonstrate that the bleeding time of suture holes after construction of arterial bypass anastomosis is shorter after treatment with Lyostypt® than with Surgicel®

DETAILED DESCRIPTION:
Hemostasis in peripheral vascular surgery is made more difficult by the need for direct arterial and arterial graft suturing as well as by systemic anticoagulation to prevent thrombosis during periods of vascular occlusion. Polytetrafluorethylene (PTFE) is one of the most frequently used graft materials for vascular replacement or bypass in the case when no autologous venae are available (1). However, the insufficient elasticity of PTFE and its porosity promote the development of suture hole bleeding (2,3) which can cause considerable loss of blood and prolongation of operations (2).

This study is designed to demonstrate the superiority of Lyostypt® to oxidized cellulose (Surgicel®) for hemostasis of suture hole bleeding in arterial bypass anastomoses after vascular reconstruction. Lyostypt® is an absorbable, wet stable collagen compress made of collagen fibrils of bovine origin. Collagen leads to thrombocyte adhesion and to activation of coagulation factor XII. Therefore collagen is very effective in hemostasis. Collagen is cell-friendly whereas other hemostats significantly disturb cell growth. Advantages of collagen fleece are fast induction of hemostasis, low tissue reaction and fast absorption (15). Furthermore, collagen was shown to be the best overall hemostatic agent in microvascular surgery. Authors concluded that collagen fleece establish faster hemostasis than oxidized cellulose and that it was resorbed faster than oxidized cellulose (15).

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for a peripheral vascular reconstruction due to peripheral vascular disease (PVD) including femoro-femoral, femoro-popliteal and femoro-crural reconstructions or the need of a crossover including femoro-femoral or ilaco-femoro reconstruction.
* suture hole bleeding of peripheral arterial bypass anastomosis using PTFE graft prosthesis
* Written informed consent

Exclusion Criteria:

* Emergency surgery
* Patients with coagulopathy or uremia
* Reoperation within one month at the same location
* Pregnant and Breastfeeding Women
* Known or suspected allergies or hypersensitivity to any of the used devices (e.g. to material of bovine origin)
* Severe comorbidity (ASA ≥ 4)
* Life expectancy less than 12 months
* Current immunosuppressive therapy (more than 40 mg of corticoid per day or ezathioprin)
* Chemotherapy within last 4 weeks
* Radiotherapy on the treated region within the last 2 months
* Severe psychiatric or neurologic diseases
* Lack of compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Time to hemostasis | Minutes

SECONDARY OUTCOMES:
Number of Complications | 30 days after surgery
Postoperative Mortality | 30 days after surgery
Efficacy Rating of Study Device evaluated by Surgeon | intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Hardy Schumacher, Prof. Dr., Study Chair — Klinikum Hanau GmbH
Locations (1):
- Klinikum Hanau GmbH, Gefaesschirurgie, Hanau, Hesse, Germany

REFERENCES:
- [Background] Bellon JM, Bujan J, Contreras LA, Hernando A, Jurado F. Similarity in behavior of polytetrafluoroethylene (ePTFE) prostheses implanted into different interfaces. J Biomed Mater Res. 1996 May;31(1):1-9. doi: 10.1002/(SICI)1097-4636(199605)31:13.0.CO;2-S. PMID 8731143
- [Background] Carney WI Jr, Lilly MP. Intraoperative evaluation of PTFE, Dacron and autogenous vein as carotid patch materials. Ann Vasc Surg. 1987 Dec;1(5):583-6. doi: 10.1016/S0890-5096(06)61445-3. PMID 2974302
- [Background] Zdrahala RJ. Small caliber vascular grafts. Part I: state of the art. J Biomater Appl. 1996 Apr;10(4):309-29. doi: 10.1177/088532829601000402. PMID 8859403
- [Background] Lumsden AB, Heyman ER; Closure Medical Surgical Sealant Study Group. Prospective randomized study evaluating an absorbable cyanoacrylate for use in vascular reconstructions. J Vasc Surg. 2006 Nov;44(5):1002-1009; discussion 1009. doi: 10.1016/j.jvs.2006.06.039. Epub 2006 Oct 3. PMID 17020801
- [Background] Miller CM, Sangiolo P, Jacobson JH 2nd. Reduced anastomotic bleeding using new sutures with a needle-suture diameter ratio of one. Surgery. 1987 Feb;101(2):156-60. PMID 3810486
- [Background] Citrin P, Doscher W, Wise L, Margolis IB. Control of needle hole bleeding with ethyl-cyanoacrylate glue (Krazy Glue). J Vasc Surg. 1985 May;2(3):488-90. doi: 10.1067/mva.1985.avs0020488. PMID 3999241
- [Background] Hait MR, Robb CA, Baxter CR, Borgmann AR, Tippett LO. Comparative evaluation of Avitene microcrystalline collagen hemostat in experimental animal wounds. Am J Surg. 1973 Mar;125(3):284-7. doi: 10.1016/0002-9610(73)90042-1. No abstract available. PMID 4570330
- [Background] Hatsuoka M, Seiki M, Sasaki K, Kashii A. Hemostatic effects of microfibrillar collagen hemostat (MCH) in experimental coagulopathy model and its mechanism of hemostasis. Thromb Res. 1986 May 1;42(3):407-12. doi: 10.1016/0049-3848(86)90269-0. No abstract available. PMID 3520941
- [Background] Silverstein ME, Keown K, Owen JA, Chvapil M. Collagen fibers as a fleece hemostatic agent. J Trauma. 1980 Aug;20(8):688-94. doi: 10.1097/00005373-198008000-00010. PMID 7401211
- [Background] Czerny M, Verrel F, Weber H, Muller N, Kircheis L, Lang W, Steckmeier B, Trubel W. Collagen patch coated with fibrin glue components. Treatment of suture hole bleedings in vascular reconstruction. J Cardiovasc Surg (Torino). 2000 Aug;41(4):553-7. PMID 11052282
- [Background] Joseph T, Adeosun A, Paes T, Bahal V. Randomised controlled trial to evaluate the efficacy of TachoComb H patches in controlling PTFE suture-hole bleeding. Eur J Vasc Endovasc Surg. 2004 May;27(5):549-52. doi: 10.1016/j.ejvs.2004.01.018. PMID 15079782
- [Background] Jackson MR, Gillespie DL, Longenecker EG, Goff JM, Fiala LA, O'Donnell SD, Gomperts ED, Navalta LA, Hestlow T, Alving BM. Hemostatic efficacy of fibrin sealant (human) on expanded poly-tetrafluoroethylene carotid patch angioplasty: a randomized clinical trial. J Vasc Surg. 1999 Sep;30(3):461-6. doi: 10.1016/s0741-5214(99)70073-x. PMID 10477639
- [Background] Taylor LM Jr, Mueller-Velten G, Koslow A, Hunter G, Naslund T, Kline R; Beriplast B Investigators. Prospective randomized multicenter trial of fibrin sealant versus thrombin-soaked gelatin sponge for suture- or needle-hole bleeding from polytetrafluoroethylene femoral artery grafts. J Vasc Surg. 2003 Oct;38(4):766-71. doi: 10.1016/s0741-5214(03)00474-9. PMID 14560228
- [Background] Glickman M, Gheissari A, Money S, Martin J, Ballard JL; CoSeal Multicenter Vascular Surgery Study Group. A polymeric sealant inhibits anastomotic suture hole bleeding more rapidly than gelfoam/thrombin: results of a randomized controlled trial. Arch Surg. 2002 Mar;137(3):326-31; discussion 332. doi: 10.1001/archsurg.137.3.326. PMID 11888460
- [Background] Schonauer C, Tessitore E, Barbagallo G, Albanese V, Moraci A. The use of local agents: bone wax, gelatin, collagen, oxidized cellulose. Eur Spine J. 2004 Oct;13 Suppl 1(Suppl 1):S89-96. doi: 10.1007/s00586-004-0727-z. Epub 2004 Jun 22. PMID 15221572
- [Background] Wachol-Drewek Z, Pfeiffer M, Scholl E. Comparative investigation of drug delivery of collagen implants saturated in antibiotic solutions and a sponge containing gentamicin. Biomaterials. 1996 Sep;17(17):1733-8. doi: 10.1016/0142-9612(96)87654-x. PMID 8866036
- [Background] Uranüs, S. ; Pfeifer, J. ; Alimoglu, O. ; Özmen, T. Laparoskopische Eingriffe an der Milz Chir Gastroenterol 2004;20(Suppl.2):35-41 (DOI:10.1159/000083352)
- [Background] Heidemann D, Hartenstein B. [Effect of local hemostyptics on human gingiva fibroblasts in culture]. Dtsch Z Mund Kiefer Gesichtschir. 1989 May-Jun;13(3):226-9. German. PMID 2625015
- [Background] Haussmann P, Mergard UE, Kohnlein HE. [Effect of various hemostatics. Animal experiment studies]. Fortschr Med. 1974 May 9;92(13):579-80. No abstract available. German. PMID 4829453
- [Background] Bauer P, Kohne K. Evaluation of experiments with adaptive interim analyses. Biometrics. 1994 Dec;50(4):1029-41. PMID 7786985
- [Background] Jensen LP, Lepantalo M, Fossdal JE, Roder OC, Jensen BS, Madsen MS, Grenager O, Fasting H, Myhre HO, Baekgaard N, Nielsen OM, Helgstrand U, Schroeder TV. Dacron or PTFE for above-knee femoropopliteal bypass. a multicenter randomised study. Eur J Vasc Endovasc Surg. 2007 Jul;34(1):44-9. doi: 10.1016/j.ejvs.2007.01.016. Epub 2007 Apr 2. PMID 17400486
- [Background] Ballotta E, Renon L, Toffano M, Da Giau G. Prospective randomized study on bilateral above-knee femoropopliteal revascularization: Polytetrafluoroethylene graft versus reversed saphenous vein. J Vasc Surg. 2003 Nov;38(5):1051-5. doi: 10.1016/s0741-5214(03)00608-6. PMID 14603216
- [Background] Devine C, McCollum C; North West Femoro-Popliteal Trial Participants. Heparin-bonded Dacron or polytetrafluorethylene for femoropopliteal bypass: five-year results of a prospective randomized multicenter clinical trial. J Vasc Surg. 2004 Nov;40(5):924-31. doi: 10.1016/j.jvs.2004.08.033. PMID 15557906
- [Background] Eiberg JP, Roder O, Stahl-Madsen M, Eldrup N, Qvarfordt P, Laursen A, Greve M, Florenes T, Nielsen OM, Seidelin C, Vestergaard-Andersen T, Schroeder TV. Fluoropolymer-coated dacron versus PTFE grafts for femorofemoral crossover bypass: randomised trial. Eur J Vasc Endovasc Surg. 2006 Oct;32(4):431-8. doi: 10.1016/j.ejvs.2006.04.018. Epub 2006 Jun 27. PMID 16807001
- [Background] Kapfer X, Meichelboeck W, Groegler FM. Comparison of carbon-impregnated and standard ePTFE prostheses in extra-anatomical anterior tibial artery bypass: a prospective randomized multicenter study. Eur J Vasc Endovasc Surg. 2006 Aug;32(2):155-68. doi: 10.1016/j.ejvs.2005.12.015. Epub 2006 Apr 17. PMID 16617028
- [Background] Klinkert P, Schepers A, Burger DH, van Bockel JH, Breslau PJ. Vein versus polytetrafluoroethylene in above-knee femoropopliteal bypass grafting: five-year results of a randomized controlled trial. J Vasc Surg. 2003 Jan;37(1):149-55. doi: 10.1067/mva.2002.86. PMID 12514593
- [Result] Qerimi B, Baumann P, Husing J, Knaebel HP, Schumacher H. Collagen hemostat significantly reduces time to hemostasis compared with cellulose: COBBANA, a single-center, randomized trial. Am J Surg. 2013 Jun;205(6):636-41. doi: 10.1016/j.amjsurg.2012.05.033. Epub 2013 Jan 17. PMID 23332688
- [Result] Baumann P, Schumacher H, Husing J, Luntz S, Knaebel HP. A randomized, controlled, prospective trial to evaluate the haemostatic effect of Lyostypt versus Surgicel in arterial bypass anastomosis: "COBBANA" trial. Trials. 2009 Sep 29;10:91. doi: 10.1186/1745-6215-10-91. PMID 19788736